CLINICAL TRIAL: NCT01269086
Title: Family Preventive Visits to Detect Risk Factors in the Family
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fundacion Hispanoamericana de Solidaridad (Unknown); Fundacion MAPFRE (Other)
Responsible Party: Diego Garcia-Huidobro, Family Medicine Department, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 00001
Record Dates: First submitted 2010-12-30; First posted 2011-01-04 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2010-10

CONDITIONS: Primary Heath Care; Preventive Medicine; Adolescent Health Services; Family; Family Practice
Keywords: Primary Heath Care; Preventive Medicine; Adolescent Health Services; Spouses; Family; Family Practice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Traditional care with no systematic assessment of family member´s health problems or risk factors.
- Family Preventive Visit (Experimental): Systematic assessment of health diseases or risk factors in the spouse and adolescent child.
  Interventions: Behavioral: Family Preventive Visit

INTERVENTIONS:
Behavioral: Family Preventive Visit — Systematic assessment of health diseases or risk factors in the spouse and adolescent child.
  Arms: Family Preventive Visit

SUMMARY:
The purpose of this study is to determine whether a systematic family assessment in adult preventive health visits increases the detection of risk factors in the spouse or adolescent child of the screened person.

ELIGIBILITY:
Inclusion Criteria:

* Parents of adolescents between 14-17 years.

Exclusion Criteria:

* Living with single parents.
* Does not accept participating in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Composite outcome: Family Risk Factors | 1 month
  The composite outcome is conformed by: detection of smoking, alcohol, substance abuse, major depression or other mental health disease, high emotional stress, suicide risk in the couple and the adolescent child; and risk of pregnancy, risk of sexually transmitted diseases, risk of eating disorders, risk of school grade repetition or school drop-out in the adolescent child, and the presence of marital or parent-child relationship problems detected by the parent/spouse.

SECONDARY OUTCOMES:
Composite outcome: Couple Risk Factors | 1 month
  The composite outcome is conformed by: detection of smoking, alcohol, substance abuse, major depression or other mental health disease, high emotional stress, suicide risk in the couple, and the presence of marital relationship problems detected by the spouse.
Composite outcome: Adolescent Risk Factors | 1 month
  The composite outcome is conformed by: smoking, alcohol, substance abuse, major depression or other mental health disease, high emotional stress, risk of suicide, risk of pregnancy, risk of sexually transmitted diseases, risk of eating disorders, risk of school grade repetition or school drop-out in the adolescent child, and the presence of parent-child relationship problems detected by the parent.
Type of health plan for follow up | 1 month
  The health plan will be categorized in comprehensive bio-psycho-social health plans or only biomedical health plans.
Diagnostic accuracy of adults to diagnose risk factors in their spouse or adolescent child. | 1 month
  We will assess sensibility, specificity, positive and negative predictive values, positive and negative likelihood ratios of parents to detect risk factors in their spouse and child.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Garcia-Huidobro, MD, Principal Investigator — Family Medicine Department, Pontificia Universidad Catolica de Chile
Locations (1):
- Centro de Salud Familiar San Alberto Hurtado, Santiago, Chile